CLINICAL TRIAL: NCT06969729
Title: Evaluation of Clinical Efficacy and Safety of Aortal Stent-graft Modelled Printing 3D Model Printing Technology - Multicenter, Randomized Clinical Trial
Brief Title: Evaluation of Clinical Efficacy and Safety of Aortal Stent-Graft Created Using 3D Printing Technology
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Samodzielny Publiczny Szpital Kliniczny nr 2 PUM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/ABM/01/00121/P/02
Record Dates: First submitted 2023-01-14; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aortic Aneurysm; Juxtarenal Aortic Aneurysm; Thoracoabdominal Aneurysm; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician-Modified Stent-Grafts Made Using 3D Aortic Template (Experimental): Patients with aortic pathology undergoing implantation of physician-modified stent-grafts created using a patient-specific 3D-printed aortic template.
  Interventions: Procedure: Physician-Modified Fenestrated Stent-Graft (3D-Printed Template-Guided)
- Custom-Made Fenestrated Stent-Graft (Active Comparator): Implantation of a commercially manufactured, patient-specific custom-made fenestrated stent-graft via an endovascular approach.
  Interventions: Procedure: Physician-Modified Fenestrated Stent-Graft (3D-Printed Template-Guided)

INTERVENTIONS:
Procedure: Physician-Modified Fenestrated Stent-Graft (3D-Printed Template-Guided) — Implantation of a physician-modified fenestrated stent-graft using a patient-specific 3D-printed aortic template, performed via an endovascular approach.

SUMMARY:
the comparison of physician-modified stent-graft created in 3D models versus custom-made devices in the treatment of complex abdominal aortic aneurysm

DETAILED DESCRIPTION:
This is randomized, multicenter, open-label, 2 -arm Study to evaluate the efficacy and safety in stent-graft application of arm A and Arm B in patients with juxtarenal or pararenal abdominal aortic aneurysm, thoracic-abdominal aneurysm type IV or type IA endoleak.

Approximately 100 eligible patients will be randomized in a 1:1 ratio into 2 arms (n=50 in each arm) Arm A treated with innovative angiosurgery intervention Arm B standard procedure Study will use an Interactive Web Response System (IWRS) for randomization. Randomization will be used to minimize bias in the assignment of subjects to treatment groups, to increase the likelihood that known and unknown subject attributes (e.g. demographic and baseline characteristics) are evenly balanced, and to enhance the validity of statistical comparisons across treatment groups.

Subjects will be randomized based on following stratification: • Site

• Aneurysm class Subject participation will include a Screening Phase, Intervention Phase, Safety follow-up and End of Study.

The screening phase will last up to 28 days before the therapeutic intervention periods starts (two hospitalizations finished with 2 angio surgery intervention) during which the subject's eligibility and baseline characteristics will be determined. The therapeutic intervention will last from randomization until second hospitalization will end with angio surgery intervention). There will be 2 follow up visits. Safety follow up will lasts 12 months.

Aorta assessment by angio CT will be performed at screening, intervention period at hospitalization no. 1 and in 30 day follow up, 12 month follow up

ELIGIBILITY:
Inclusion Criteria:

Female and male subjects age ≥ 18 2. Subject need to meet one of the following criteria:

* Subjects with juxtarenal or suprarenal abdominal aortic aneurysm, type IV thoracoabdominal aneurysm of diameter >5.5cm (male) and 5.2cm (female)
* Subjects with juxtarenal or suprarenal abdominal aortic aneurysm, type IV thoraco-abdominal aneurysm with aneurysm growth rate ≥ 0.5cm during 6 months
* Type IA endoleak of post-implantation of abdominal stent- graft 3. Iliac arteries morphology with aortic stent graft implantation to be restored 4. Aortic segment which is proximal to aneurysm
* Length ≥20mm
* Diameter 20mm-36mm
* Aortic suprarenal angle ≤75 degrees 5. Survival > 2 years

Exclusion Criteria:

1. Female and male subjects age <18
2. Pregnancy and breast feeding
3. Allergy and hypersensitivity to matherials of which the stent- graft is composed
4. Hypersensitivity and contraindication to anti coagulation or contrast application to angio - CT which cannot be eliminated medically
5. Coagulopathy which cannot medically treated
6. Active infection which might cause stent - graft infection
7. Creatinine level > 3.0mg/dL
8. Marphan syndrome, Ehlers - Denlos syndrome
9. Unstable angina pectoris
10. Raptured aortic aneurysm caused by cardiac insufficiency
11. Unwillingness to comply with protocol procedures
12. Iliac arteries morphology adequate for stent-graft implantation
13. The diameter of the aortic flow lumen in reno-visceral aorta greater than 34mm
14. Aortic section which is proximal to celiac artery with significant number of thrombi, calcification or changed by aneurysm
15. Aorta with significant number of irregular thrombi which may lead to embolism ("shaggy aorta")
16. Diameter of proximal kidney arteries which is exercisable to stenting <4.5mm
17. Devision of kidney artery which is exercisable to stenting in the distance of <1cm of celiac artery, each of them is is in <4.5mm in diameter
18. Atypical anatomy of celiac artery in the form of separate exit of splenic and hepatic aortic artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Surviving at 1 Year Without Aortic Rupture | 1 year
  Rupture - free one year survival. The number of participants who remain alive and free from aortic rupture at 1 year following stent-graft implantation. Rupture will be defined as radiologically confirmed loss of aortic wall integrity with associated clinical symptoms.
Number of Participants Surviving at 30 Days Post-Procedure (Perioperative Survival) | 30 days
  The number of participants who are alive 30 days after the stent-graft procedure. Deaths from any cause within 30 days post-implantation will be counted.

SECONDARY OUTCOMES:
Number of Deaths from Any Cause Within 1 Year | 1 year
  Total number of participant deaths due to any cause occurring within one year of the procedure.
Number of Cardiovascular-Related Deaths Within 1 Year | 1 year
  The number of participant deaths attributed to cardiovascular causes (e.g., myocardial infarction, stroke, aortic rupture) within 1 year of the procedure, as adjudicated by the study investigators.
Number of Participants Without Aneurysm Growth at 1 Year | 1 year
  The number of participants whose aneurysm size remains stable (no increase >5 mm in maximum diameter) as assessed by imaging (e.g., CT angiography) at 1 year post-implantation.
Number of Participants Surviving Without Reintervention at 1 Year | 1 year
  The number of participants who do not require any secondary endovascular or surgical intervention related to the index aortic pathology within 1 year of the initial procedure.
Change in Incidence of Cardiovascular Events at 1 Year | 1 year
  Change in the number of participants experiencing cardiovascular events (e.g., myocardial infarction, stroke, cardiac arrest) compared to baseline rates or historical controls over a 1-year follow-up period.
Number of Deaths from Any Cause at 1 Year (Overall Mortality) | 1 year
  The total number of participant deaths from any cause within one year of the stent-graft procedure.
Change in Renal Function at 1 Year | 1 year
  Change in estimated glomerular filtration rate (eGFR) or serum creatinine level from baseline to 1 year post-procedure, used to assess renal function.
Total Cost of Treatment at 1 Year | 1 year
  Cumulative healthcare cost per participant associated with the initial stent-graft procedure, hospitalization, follow-up visits, imaging, medications, and any reinterventions within 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- An Independent Clinical Hospital 2 PUM, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional data governance policies and applicable data protection regulations, including the General Data Protection Regulation (GDPR) and national laws. These frameworks restrict the sharing of detailed clinical data with external parties to ensure the confidentiality and security of participant information.